CLINICAL TRIAL: NCT07167524
Title: Evaluation of the Dialytic Clearance of the Combination of Peracillin and Tazobactam in Patients Receiving Continuous Renal Replacement Therapy in Intensive Care
Brief Title: Evaluation of the Dialytic Clearance of the Combination of Peracillin and Tazobactam
Acronym: EPIC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0306/OB; 2025-A00885-44 (Other: ANSM)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Severe Bacterial Infections
Keywords: medical resuscitation; antibiotic therapy; clearance of piperacillin and tazobactam
MeSH Terms: conditions — Sepsis; Bacterial Infections | interventions — Tazobactam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected at baseline, T15min, T30min, T45min, T1h, T3h, T6h, T8h, T12h, T24h, T36h in pre-filter (before pre-dilution when present), post-filter (after post-dilution when present), in the effluent and in the urine in case of preserved diuresis.
  Biological samples will be collected in EDTA tubes with a capacity of 2mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Dosage concentration of piperacillin and tazobactam — The concentration of piperacillin and tazobactam will be quantified by liquid chromatography coupled with tandem mass spectrometry (HPLC-MS² - CIC-CRB 1404) at each of these times by transposition of the method already used in current practice.

SUMMARY:
Severe bacterial infections, often responsible for sepsis and septic shock, are a major challenge in critical care: approximately 50% of patients are affected, with a mortality rate of up to 40%. Their initial management consists of antibiotic therapy with an adapted spectrum of activity and dose. One of the most widely used antibiotic therapies in intensive care is the piperacillin-tazobactam (pip-taz) combination, a beta-lactam combined with a beta-lactamase inhibitor, which is indicated probabilistically in many infections (pneumopathies, intra-abdominal infections, urinary tract infections, etc.). Mortality rates of up to 40%. Their initial management consists of antibiotic therapy with an appropriate spectrum of activity and dose. One of the most widely used antibiotic therapies in intensive care is the piperacillin-tazobactam (pip-taz) combination, a beta-lactam combined with a beta-lactamase inhibitor, which is indicated probabilistically in many infections (pneumonia, intra-abdominal infections, urinary tract infections, etc.).

Intensive care patients with septic shock exhibit specific pharmacokinetics with an increased volume of distribution, notably due to significant capillary leakage, often disrupted hepatic metabolism, possible hypoalbuminemia, the presence of renal hyperclearance in the initial phase or conversely, the onset of renal failure with altered glomerular filtration rate, sometimes leading to extrarenal clearance, changes that have consequences for the efficacy and toxicity of the administered antibiotic therapy. Sepsis itself also causes renal dysfunction, with the main pathophysiological hypotheses being an alteration of microcirculation, cellular metabolic reprogramming, and deregulation of the inflammatory response. It is therefore essential to focus on the dosages administered and the pharmacokinetics of these patients. Indeed, underdosing is associated with the emergence of resistance and a poorer prognosis in intensive care patients: increased risk of treatment failure, length of stay and mortality. Conversely, significant overdoses can be associated with a poorer renal prognosis, seizures, encephalopathy which can lead to delayed awakening, prolonged duration of mechanical ventilation and intensive care stay.

DETAILED DESCRIPTION:
Pip-taz is administered intravenously due to non-absorption via the oral route. It is weakly bound to plasma proteins (21%), inducing good clearance of extrarenal clearance (fraction extracted in 4 hours: 23.6% of the administered dose). Its plasma half-life is 60 minutes. This molecule is not metabolized, and is therefore independent of liver function. It is eliminated mainly in active form in the urine (65%) and bile (35%). Thus, the main determinant of pip-taz clearance is renal clearance, or continuous extrarenal clearance (CER) in dialysis patients in intensive care.

Pip-taz is characterized by time-dependent pharmacodynamics, with better coverage with continuous infusions compared to discontinuous infusions. However, there is no well-defined pattern in patients undergoing continuous extra-renal purification. Despite recommendations regarding antibiotic dosages for use in intensive care, the lack of data regarding patients undergoing continuous renal replacement therapy (CRRE) remains a major and complex problem in optimizing treatment, as these patients present with unique pharmacokinetics, with an increased risk of treatment failure and mortality. Furthermore, there has been a change in practices in recent years, with pip-taz being administered by continuous infusion and increasingly less by discontinuous infusion, in accordance with the latest recommendations.

To our knowledge, few studies have examined the pharmacokinetics of the pip-taz combination in patients undergoing cCRRE in intensive care. Most of these rare studies did not use standard pip-taz dosages, did not examine the clinical and biological variables influencing pip-taz clearance, and none have examined the impact of any preserved diuresis. Furthermore, there are no data on the kinetics of tazobactam in this population. It therefore seems relevant, given the frequent use of this antibiotic therapy in patients undergoing cERE, to accurately assess the clearance of piperacillin and tazobactam in this population. From a precision medicine perspective, these data could contribute to the construction of a pharmacokinetic model using a population approach, based on blood, urine, and effluent samples, in order to provide a tool to assist in the prescription of this antibiotic therapy in intensive care to reduce iatrogenicity and optimize its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age;
* Patient admitted to intensive care with a prescription for cREV (CVVH (pre- or post-dilution (convection)), CVVHD (diffusion), CVVHDF);
* Diagnosed or suspected infection sensitive to the piperacillin-tazobactam combination administered by continuous infusion as part of the patient's standard care;
* Concomitant prescription of piperacillin-tazobactam and cREV;
* Patient affiliated with a social security scheme;
* Adult who has read and understood the information letter and has not expressed non-opposition. Due to the potential life-threatening emergency, if the patient is unable to express their non-opposition, the consent of a trusted person or, where applicable, relatives will be sought.

Exclusion Criteria:

* Documented or suspected allergy to penicillins;
* Opposition from the patient or trusted person;
* Pregnant, childbirth, or breastfeeding woman;
* Minor patient;
* Person deprived of liberty by an administrative or judicial decision;
* Person placed under judicial protection, guardianship, or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing continuous extra-renal purification (CER) in the various intensive care units of the Rouen University Hospital (surgical, medical, cardiac surgical), receiving concomitant antibiotic therapy with piperacillin-tazobactam (initiated before or after CER) for sepsis or septic shock.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Determination of continuous extrarenal clearance (CERC) of piperacillin in patients with infection in intensive care | At Enrollment visit, Time 15 minutes, 30 minutes and 45 minutes, Time 1 hour, 3 hours, 6 hours, 8 hours, 12 hours, 24 hours and 36 hours in pre-filter (before pre-dilution when present), post-filter (after post-dilution when present)
  The cERC clearance of piperacillin will depend on the type of cERC used, thus determining a clearance:
  * diffusion (dialysis, continuous venomous hemodialysis (CVVHD)),
  * convection (filtration, continuous venomous hemofiltration (CVVH)),
  * diffusion and convection (dialysis and filtration, continuous venomous hemodiafiltration (CVVHDF)).
  Each of these clearances will be characterized by different formulas, based on the collection of the following parameters: pre- and post-filter concentrations, concentration in the dialysate/filtrate/effluent, cERC flow rate for diffusion and convection, hematocrit, and partition coefficient of the substance between whole blood and plasma.

SECONDARY OUTCOMES:
Determination of EERc clearance of tazobactam | At Enrollment visit, Time 15 minutes, 30 minutes and 45 minutes, Time 1 hour, 3 hours, 6 hours, 8 hours, 12 hours, 24 hours and 36 hours in pre-filter (before pre-dilution when present), post-filter (after post-dilution when present)
  The cERC clearance of tazobactam will depend on the type of cERC used, thus determining a clearance: - diffusion (dialysis, continuous venomous hemodialysis (CVVHD)), - convection (filtration, continuous venomous hemofiltration (CVVH)), - diffusion and convection (dialysis and filtration, continuous venomous hemodiafiltration (CVVHDF)). Each of these clearances will be characterized by different formulas, based on the collection of the following parameters: pre- and post-filter concentrations, concentration in the dialysate/filtrate/effluent, cERC flow rate for diffusion and convection, hematocrit, and partition coefficient of the substance between whole blood and plasma.
Evaluation of total clearance of piperacillin in patients with preserved residual diuresis. | At Enrollment visit, Time 15 minutes, 30 minutes and 45 minutes, Time 1 hour, 3 hours, 6 hours, 8 hours, 12 hours, 24 hours and 36 hours in pre-filter (before pre-dilution when present), post-filter (after post-dilution when present)
  The total clearance (CLT) of piperacillin will be determined by considering that they correspond to the sum of the renal clearance (CLR) and the clearance of the EERc (CLEERc). Thus, CLT = CLR + CLEERc. In the absence of diuresis, CLR=0 will be considered and therefore CLT = CLEERc.
Evaluation of total clearance of tazobactam in patients with preserved residual diuresis. | At Enrollment visit, Time 15 minutes, 30 minutes and 45 minutes, Time 1 hour, 3 hours, 6 hours, 8 hours, 12 hours, 24 hours and 36 hours in pre-filter (before pre-dilution when present), post-filter (after post-dilution when present)
  The total clearance (CLT) of tazobactam will be determined by considering that they correspond to the sum of the renal clearance (CLR) and the clearance of the EERc (CLEERc). Thus, CLT = CLR + CLEERc. In the absence of diuresis, CLR=0 will be considered and therefore CLT = CLEERc.
Description of the evolution of plasma concentrations of piperacillin over time. | At 36 hours
  Plasma concentrations of piperacillin over time will be evaluated using a population pharmacokinetic model using a nonlinear mixed-effects regression model.
Description of the evolution of plasma concentrations of tazobactam over time. | At 36 hours
  Plasma concentrations of tazobactam over time will be evaluated using a population pharmacokinetic model using a nonlinear mixed-effects regression model.
Development of a dosage regimen to optimize the benefit/risk balance | At 36 hours
  A dosage regimen to optimize the benefit/risk balance in this population will be developed by plotting the probability curves of reaching the therapeutic target (PTA) as a function of increasing MICs. The pharmacodynamic indices of efficacy retained will be the fraction of time where the free piperacillin concentration is greater than 1x the MIC (fT > 1xMIC = 100%) and 4x the MIC (fT > 4xMIC = 100%).

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.